CLINICAL TRIAL: NCT01536509
Title: Telehealth Enhancement of Adherence to Medication in Pediatric Inflammatory Bowel Disease
Brief Title: Improving Medication Adherence in Pediatric Inflammatory Bowel Disease
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD067174 (NIH)
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telehealth Behavioral Treatment (Experimental)
  Interventions: Behavioral: Telehealth Behavioral Treatment (TBT)
- Education Only (Active Comparator)
  Interventions: Behavioral: Education Only (EO)

INTERVENTIONS:
Behavioral: Telehealth Behavioral Treatment (TBT) — Families in the TBT condition will receive three individually-tailored behavioral intervention sessions in addition to the online education intervention with 1) guided problem-solving and behavior management training tailored to the unique needs and/or barriers of the family, and 2) discussion of the patient's adherence since the previous session. In addition, patients in the TBT condition will be signed up for text message reminder service offered free of charge via www.mymedschedule.com. These are generic reminder text messages are used to assist with adherence in adolescents. Intervention sessions will be conducted via telehealth delivery with trained postdoctoral psychology fellows or masters-level graduates using webcams, supplied by the study, and SkypeTM free software.
  Arms: Telehealth Behavioral Treatment
Behavioral: Education Only (EO) — Families in the EO condition will receive three individual sessions in addition to the online education intervention to review 1) online educational intervention material to answer questions participants have, 2) educational brochures from the Crohn's and Colitis Foundation of America (CCFA), which contain additional information (e.g., Guide for Parents, Living with IBD, Guide for Kids and Teenagers), and 3) general healthy lifestyle recommendations (e.g., sleep, exercise, etc.). Sessions will be conducted via telehealth delivery with trained postdoctoral clinical psychology fellows or masters-level graduates using webcams, supplied by the study, and SkypeTM free software.
  Arms: Education Only

SUMMARY:
The purpose of the study is to test an online behavioral intervention to improve medication adherence in children diagnosed with Inflammatory Bowel Disease. Interested families will be monitored for four weeks to determine how frequently their child's IBD medication is taken. Patient's taking less than 90% of medications will be randomized to one of two intervention conditions to complete intervention sessions online. The study consists of 4 online intervention sessions with topics differing by condition and 5 online assessments to complete quality of life questionnaires over a 14 month time frame.

DETAILED DESCRIPTION:
The purpose of the study is to test the efficacy of a telehealth behavioral treatment (TBT) protocol to improve medication adherence in children and adolescents with IBD via a randomized controlled clinical trial. Participants in the TBT condition will be compared to those in an education only (EO) condition. In order to examine clinical significance of the intervention, treatment outcomes will include disease severity, HRQOL, and health care utilization. This randomized controlled clinical trial for nonadherence to medication randomizes participants to either the TBT or EO intervention condition, with assessments occurring at baseline, post-treatment, and 3-, 6-, and 12-month follow-up. Both conditions will participate in a self-guided educational intervention during week 6 of enrollment, with three intervention sessions at weeks 8, 10, and 12. A 4-week run-in phase immediately preceding randomization is utilized to establish participants' baseline adherence. Assessments will occur at week 5 (Baseline Assessment 1), week 14 (Post-treatment Assessment 2), and 3-, 6-, and 12-month post-treatment follow-up (Assessments 3, 4, and 5). Intervention topics will differ for each condition; however, the frequency of contact is equivalent across conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently seen for care at one of the collaborating research sites: Cincinnati Children's Hospital Medical Center, Connecticut Children's Medical Center, Children's Hospital of Philadelphia, Nationwide Children's Hospital, University of California San Francisco Benioff Children's Hospital, or Children's Mercy Hospitals and Clinics
* Patient diagnosed with Crohn's disease, ulcerative colitis, or indeterminate colitis
* Patient age between 11-18 years
* Patient currently living at home
* Patient currently prescribed at least one daily oral immunomodulator (e.g., 6-MP/azathioprine) and/or 5-ASA (e.g., mesalamine)in pill form
* English fluency for patient and parents
* Inclusion for Randomization: <90% adherence to immunomodulator and/or 5-ASA during four week run-in phase

Exclusion Criteria:

* Diagnosis of pervasive developmental disorder in patient or parent
* Diagnosis of serious mental illness (e.g., schizophrenia) in patient or parent

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2012-02; Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 15 months
  Medication adherence will be measured using electronic monitoring. The specific device is the MEMS TrackCap. Immunomodulators and/or mesalamine medications will be assessed.

SECONDARY OUTCOMES:
Health-related quality of life | 15 months
  The IMPACT III measure will be used for this assessment. This is an IBD-specific HRQOL assessment tool.
Disease Severity | 15 months
  The Pediatric Crohn's Disease Activity Index (PCDAI) and Partial Harvey-Bradshaw Index (PHBI) will be used to assess disease severity in patients with Crohn's disease. The Pediatric Ulcerative Colitis Index (PUCAI) will be used in patients with ulcerative colitis.
Health care utilization | 15 months
  Health care utilization will be assessed via medical chart review and all IBD-related hospital admissions, procedures, communications, clinic appointments, and other encounters with the health care system will serve as indicators of utilization.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hommel, Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati; Robert Baldassano, M.D., Study Chair — Children's Hospital of Philadelphia; Wallace Crandall, M.D., Study Chair — Nationwide Children's Hospital; Francisco Sylvester, M.D., Study Chair — Connecticut Children's Medical Center; Lee Denson, M.D., Study Chair — Children's Hospital Medical Center, Cincinnati; Michele Maddux, Ph.D., Study Chair — Children's Mercy Hospital Kansas City; Melvin Heyman, M.D., Study Chair — University of California San Francisco Benioff Children's Hospital; David Keljo, M.D., Study Chair — University of Pittsburgh
Locations (9):
- United States (9):
  - University of California San Francisco Benioff Children's Hospital, San Francisco, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oklahoma State University, Stillwater, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391